CLINICAL TRIAL: NCT04730596
Title: The Effect of Ketamine and Dexmedetomidine on the Postoperative Cognitive Dysfunction After Cataract Surgery: Randomized Controlled Double-blinded Study
Brief Title: Cognitive Dysfunction After Cataract Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Collaborators: Magrabi Hospital - Doha (Unknown)
Responsible Party: Principal Investigator, Mohamed Elsayed Oriby, Lecture of Anesthesia and Intensive Care - faculty of Medicine, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: MEEC-IRB- 2021-102
Record Dates: First submitted 2021-01-26; First posted 2021-01-29 (Actual); Last update posted 2021-04-20 (Actual); Status verified 2021-04

CONDITIONS: POCD - Postoperative Cognitive Dysfunction
Keywords: Ketamine; Dexmedetomidine; cataract; Cognitive dysfunction
MeSH Terms: conditions — Postoperative Cognitive Complications; Cataract; Cognitive Dysfunction | interventions — Ketamine; Dexmedetomidine; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: * The patients will be blinded to their groups.
  * An anesthesia resident who will not participate in the study and have no the subsequent rule in it will help in the preparation of local anesthetic mixtures under strict aseptic precautions.
  * An assistant nurse who will be blinded to the study groups and will have no the subsequent rule in it will help in the collection of the data of measurements
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group I (Control group) (Placebo Comparator): - The patients in this group will receive normal saline in a labeled syringe which will be prepared by an assistant nurse not participating in the study.
  Interventions: Drug: Normal saline
- Group II (Ketamine group) (Experimental): - The patients in this group will receive ketamine at a dose of 0.3 mg/kg dissolved in normal saline in a labeled syringe which will be prepared by an assistant nurse not participating in the study.
  Interventions: Drug: Ketamine
- Group III (Dexmedetomidine group) (Experimental): - The patients in this group will receive Dexmedetomidine in a dose of 0.5 ug/kg dissolved in normal saline in a labeled syringe which will be prepared by an assistant nurse not participating in the study.
  Interventions: Drug: Dexmedetomidine

INTERVENTIONS:
Drug: Ketamine — Ketamine at a dose of 0.3 mg/kg dissolved in normal saline.
  Arms: Group II (Ketamine group)
Drug: Dexmedetomidine — Dexmedetomidine at a dose of 0.5 ug/kg dissolved in normal saline.
  Arms: Group III (Dexmedetomidine group)
Drug: Normal saline — Normal saline in a labeled syringe
  Arms: Group I (Control group)

SUMMARY:
* Cataract surgery is commonly performed in elderly patients who are at high risk for developing postoperative cognitive dysfunction. Most cataract surgeries are performed under peribulbar or retrobulbar anesthesia, however, most of the patients require sedation to relieve the perioperative anxiety and induce amnesia. So, many sedative agents can be used especially benzodiazepines which may increase the risk of developing postoperative cognitive dysfunction.
* Ketamine can be used as a sedative and analgesic agent in a dose of 0.25 -0.5 mg/kg with certain studies suggesting that it may decrease the risk of postoperative cognitive dysfunction. Similarly, dexmedetomidine can be used as a sedative and analgesic agent with the possibility of decreasing the incidence of postoperative cognitive dysfunction.
* this controlled study will compare the effect of ketamine or dexmedetomidine on the POCD of patients undergoing cataract surgery.

DETAILED DESCRIPTION:
* Postoperative cognitive dysfunction is a common postoperative complication in elderly patients. Despite the role of the risk of anesthesia and/or surgery in developing postoperative cognitive dysfunction, it can be developed even with surgeries performed under local or regional anesthesia.
* Ageing is the most common risk factor for developing postoperative cognitive dysfunction that can affect memory and speech. Also, impaired vision may be another important risk factor.
* Cataract surgeries can be considered the most common surgery performed in elderly patients. It is usually performed under local anesthesia (peribulbar, retrobulbar, or sub-tenon blocks), however, sedation is usually required to relieve the anxiety of the patients and induce amnesia.
* there are many sedative agents that can be used with such patients, the most commonly used are benzodiazepines. However, benzodiazepines use may increase the incidence of postoperative cognitive dysfunction.
* Ketamine, the dissociative anesthetic, acts mainly through inhibition of NMDA receptors that reduce the neuronal loss of the cortex. it may attenuate the postoperative cognitive dysfunction and induce neuroprotective effect through suppressing the inflammatory response and minimizing cerebral ischemia.
* dexmedetomidine is a sedative and analgesic agent that have the advantage of minimal respiratory depression and can be used as a sedative agent in cataract surgery. Studied revealed that its sedative analgesic effect is not associated with changes in memory.
* This randomized controlled double-blinded study will be carried upon 90 elderly patients undergoing cataract surgery under peribulbar anesthesia where they will be classified into 3 groups: - Group I (Placebo Group). Where the patients will receive normal saline as a placebo.

Group II (Ketamine group). Where patients will receive ketamine in a dose of 0.3 mg/kg in physiological solution.

Group III (Dexmedetomidine group). where patients will receive dexmedetomidine in a dose of 0.5 ug/kg in a physiological solution.

-Primary outcome will be the incidence of POCD, the secondary outcomes will be the hemodynamic changes and the changes in the intraocular pressure.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 65 years presented for cataract surgery under peribulbar anesthesia.

Exclusion Criteria:

* Patients with a history of psychological disorders as psychosis, schizophrenia, nephropathy.
* Patients with uncontrolled medical conditions as D.M and hypertension.
* Known allergy to the used medications
* patients with hepatic, renal, or heart failure
* Patients receiving anti-psychotic or anti-depressant medications.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

PRIMARY OUTCOMES:
The postoperative cognitive function | Within the first 3 days after surgery
  Short Portable Mental Status Questionnaire (SPMSQ) It is a score system that depends upon the number of errors in 10 questions asked to the patient where; - 0-2 errors: normal mental functioning
  3-4 errors: mild cognitive impairment
  5-7 errors: moderate cognitive impairment
  8 or more errors: severe cognitive impairment Mental Status Questionnaire (SPMSQ) score will be used to assess the cognitive dysfunction

SECONDARY OUTCOMES:
Change in the intraocular pressure | Throughout the whole intraoperative period
  The IOP will be measured before the peribulbar anesthesia, min, 5 min and 10 min after peribulbar injection, then immediately after surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Oreby, M.D, Principal Investigator — Tanta University
Locations (1):
- Faculty of Medicine, Tanta, Algharbia Governate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data of the primary outcome will be available with the corresponding author till 6 months after approval of the publication of the trial.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: till 6 months after approval of the publication of the trial.
Access Criteria: Contact the principle investigator